CLINICAL TRIAL: NCT05385094
Title: Consistency Between Measures of Renal Function in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, Associate Profesor, Senior Consultant, Karolinska University Hospital
Other Study IDs: EPN 2017/806-31 Renal Function
Record Dates: First submitted 2021-12-12; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: S Creatinine concentration
Diagnostic Test: Serum Cystatin C concentration
Diagnostic Test: Urinary Creatinine Clearance

SUMMARY:
This study aim to compare different measures of renal function (glomerular filtration rate) in ICU patients.

DETAILED DESCRIPTION:
The study uses a large dataset of prospectively collected data according to clinical routines.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with at least one measurement of urinary creatinine clearance

Exclusion Criteria:

* Renal replacement therapy initiated before the measurement of creatinine clerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlations between estimates of renal function | 7 days
Correlations between changes in estimates of renal function | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
No plan.